CLINICAL TRIAL: NCT00253955
Title: An Open-Label, Multicenter, Multinational, Centrally Randomized, Two-Arm Parallel-Group Study to Demonstrate the Non-Inferiority in Clinical Efficacy of Levofloxacin 750mg od in Comparison With Piperacillin/Tazobactam 4g/500mg Every 8 Hours in the Treatment of Mild to Moderate Hospital-Acquired Pneumonia Adult Patients in Both General Wards and ICU (Intensive Care Unit)
Brief Title: Study to Demonstrate the Clinical Efficacy of Levofloxacin in the Treatment of Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR355_3035
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2008-11-10 (Estimated); Status verified 2008-11

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Levofloxacin; Piperacillin, Tazobactam Drug Combination

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Levofloxacin
- 2 (Active Comparator)
  Interventions: Drug: Piperacillin/Tazobactam

INTERVENTIONS:
Drug: Levofloxacin
  Arms: 1
Drug: Piperacillin/Tazobactam
  Arms: 2

SUMMARY:
Primary Objective:

* The primary objective of the study is to demonstrate the non-inferiority in clinical efficacy at the test of cure (TOC) visit planned 5-7 days after treatment completion of levofloxacin 750 mg once daily (od) in comparison with piperacillin/tazobactam 4 g/500 mg every 8 hours in treating adult patients suffering from mild to moderate hospital-acquired pneumonia.

Secondary Objectives:

The secondary objectives of the study are:

* To assess the bacteriological efficacy at the test of cure (TOC) visit
* To assess the clinical and bacteriological efficacy at the end of study (EOS) visit, 28 to 32 days after treatment ends
* To assess the tolerability of both drugs

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria will be considered for enrollment into the study:

* General ward or ICU hospitalized subject.
* Subject with diagnosis of hospital-acquired pneumonia of presumed bacterial origin based upon:

  * Infection developing after at least 72 hours following hospital admission and
  * At least three of the four following signs:

    * Fever, defined as body temperature (oral or tympanic temperature ≥ 38°C or rectal temperature ≥ 38.5°C)
    * Purulent tracheal sputum production/secretion or change in sputum character
    * Total peripheral white blood cell (WBC) count > 12 G/L or < 4.5 G/L or 15% immature neutrophils (bands), regardless of total peripheral WBC count
    * Increased plasma or serum C reactive protein (CRP) level as shown by a level of at least twice the upper boundary of the hospital normal range and
    * Chest X-ray findings (anterior posterior [AP] or posterior anterior [PA], if possible lateral view) in agreement with the clinical diagnosis of bacterial pneumonia, i.e. appearance of new, progressive pulmonary infiltrate(s) attributable to infectious etiology.
* Subjects are required to have specimens collected for microbiological documentation within 24 hours prior to enrolment. Specimens should include at least one invasive or noninvasive lower respiratory tract specimen for Gram stain, culture and susceptibility testing, and at least 2 venous blood samples for culture and susceptibility testing.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

Related to the hospital-acquired pneumonia (HAP):

* Suspected viral or fungal pneumonia, or HAP strongly suspected to be caused by MRSA (methicillin-resistant Staphylococcus aureus) or organisms responsible for atypical pneumonia, such as Chlamydia pneumoniae, Legionella pneumophila or Mycoplasma pneumoniae
* Patients with severe HAP, defined as presence of at least one of the following:

  * In previously non-ventilated patients: need for mechanical ventilation consequently to HAP
  * In previously ventilated patients: oxygenation rate defined by partial pressure of oxygen in arterial blood (PaO2)/fraction of inspired oxygen (FiO2) < 200
* Radiographic findings compatible with severe HAP, i.e. showing either:

  * Rapid progression (e.g. increase in the size of the opacity by ≥ 50% within 48 hours of the current evaluation)
  * OR multilobar pneumonia (> 2 lobes) or involvement of both lungs
  * OR cavitation of a lung infiltrate
* Evidence of severe sepsis with hypotension and/or end-organ dysfunction, i.e.:

  * Shock commonly evidenced by: systolic blood pressure < 90 mmHg or diastolic blood pressure < 60 mmHg
  * In absence of previous vasopressors use, vasopressors use (except for fluid replacement) for more than 4 hours
  * In presence of vasopressors use, increase in vasopressors use (except for fluid replacement) for more than 4 hours
  * OR marked reduction in urine output (unless another explanation is available), i.e. in 1 hour: < 20 mL or in 4 hours: < 80 mL
  * OR acute renal failure requiring dialysis
  * OR profound alteration of mental status, i.e. marked lethargy/stupor/coma

Related to medical history/concomitant conditions:

* Patients with any concomitant pulmonary diseases, conditions or complications that could confound the interpretation or evaluation of drug efficacy or safety, including severe bronchiectases, cystic fibrosis, active pulmonary tuberculosis or acute pulmonary embolism, empyema, lung abscess or extra pulmonary extension of the LRTI (lower respiratory tract infection), such as meningitis, septic arthritis, endocarditis, known bronchial obstruction due to tumor or foreign body or with a history of post-obstructive pneumonia (this does not exclude patients with COPD [chronic obstructive pulmonary disease]), primary lung cancer or another malignancy metastatic to the lungs, and/or requiring chemotherapeutic treatment (for this or other reasons)
* Patients with any known or suspected bacterial infection other than the disease under investigation which will require concomitant use of a systemic antimicrobial agent other than the study drug allocated
* Patients who have received previous systemic antibiotics longer than 24 hours within 72 hours prior to the enrolment for the same episode of HAP
* Body weight > 95 kg
* Patients with impaired renal function, as shown by creatinine clearance < 20 mL/min
* Hepatic cirrhosis with Child-Pugh score > or = B
* Immuno-compromised patients, such as those presenting with either:

  * Known HIV infection with a CD4 + T-lymphocyte count < 0.2 G/L (i.e. < 200 cells/mm3)
  * Neutropenia - neutrophil count < 1.0 G/I (i.e. < 1000/mm3)
  * Patients on maintenance (≥ 3 months) corticosteroid therapy (> 20 mg/day equivalent prednisolone)

Related to study drugs:

* Patients with a microbiologically documented infection with a pathogen known prior to inclusion to be resistant to at least one of the study medications
* Patients with known or suspected hypersensitivity to, or known or suspected serious adverse reaction to levofloxacin and/or piperacillin/tazobactam and/or any other quinolones, beta-lactamase inhibitors, penicillins and/or to cephalosporins
* Patients with epilepsy or a history of epilepsy or with predisposition to seizures (e.g. patients with pre-existing central nervous system lesions)
* Patients with known or suspected history of tendon disorders unless a potential relationship to fluoroquinolone administration has been excluded.
* Patients with latent or actual known defects in glucose-6-phosphate dehydrogenase activity

General:

* Women who are breast-feeding, or are failing to use adequate contraception; for example, systemic hormones (birth control pills, implant), intrauterine device or barrier method (diaphragm with intravaginal spermicide, cervical cap, male or female condom), or are pregnant, as demonstrated by urine or serum pregnancy tests carried out before exposure to study medication or the start of any study procedure that could pose a risk to the foetus
* Patients with a recent (within three months prior to study entry) history of drug or alcohol abuse
* Patients who have received any investigational drug within one month prior to study entry.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2003-06; Primary Completion 2007-05 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy data:-Infection related signs and symptoms-Chest X-ray | from the start to the end of the study

SECONDARY OUTCOMES:
Safety data: Clinical adverse event reporting, including SAE reporting | From the inform consent signed until the end of the study
Bacteriological efficacy data:-Cultures and susceptibility testing | from the start to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Perdriset, Study Director — Sanofi
Locations (17):
- Sanofi-Aventis, Vienna, Austria
- Sanofi-Aventis, Brussels, Belgium
- Sanofi-Aventis, Prague, Czechia
- Sanofi-Aventis, Paris, France
- Sanofi-Aventis, Berlin, Germany
- Sanofi-Aventis, Athens, Greece
- Sanofi-Aventis, Guatemala City, Guatemala
- Sanofi-Aventis, Milan, Italy
- Sanofi-Aventis, Beirut, Lebanon
- Sanofi-Aventis, México, Mexico
- Sanofi-Aventis, Gouda, Netherlands
- Sanofi-Aventis, Bucharest, Romania
- Sanofi-Aventis, Moscow, Russia
- Sanofi-Aventis, Johannesburg, South Africa
- Sanofi-Aventis, Barcelona, Spain
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis, Caracas, Venezuela